CLINICAL TRIAL: NCT02413021
Title: Phase 1 Study of Deferasirox in Acute Leukemia Patients Not Treated by Standard Chemotherapy Regimens
Brief Title: The Effect of Deferasirox on Response Rate of Acute Leukemia Patients Not Treated by Standard Chemotherapy Regimens
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Golnaz Vaseghi, Dr, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78001
Record Dates: First submitted 2015-01-10; First posted 2015-04-09 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia
Keywords: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; deferasirox
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deferasirox + cytarabine (Experimental): deferasirox + cytarabine group will receive oral deferasirox at 20 mg/kg per day and cytarabine at20 mg/m^2 , SC , two times a day for 10 days every 30 days for 1 cycle.
  Interventions: Drug: Cytarabine; Drug: Deferasirox
- cytarabine (Active Comparator): cytarabine group will receive just cytarabine at 20 mg/m^2 , SC , two times a day for 10 days every 30 days for 1 cycle.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — 20 mg/m^2 , SC, two times a day for 10 days every 30 days for 1 cycle
  Other Names: Cytosar
Drug: Deferasirox — 20 mg/kg ,oral, per day
  Other Names: osveral
  Arms: deferasirox + cytarabine

SUMMARY:
The purpose of this study is to determine whether deferasirox is effective in the treatment of acute lymphatic leukemia (ALL) and acute Myeloid leukemia (AML).

DETAILED DESCRIPTION:
Many studies have demonstrated that Iron is essential for the metabolism, cell cycle regulation and metastasis in different cancer cell lines. It is also believed that Iron concentration will increase in cancer cells by enhancing expression of TFR-1 receptors and in case of receptor saturation, non-receptor-mediated pinocytosis would be a significant pathway for more iron intake. Iron deficiency may lead to increase P 53 which consequently will stop cell mitosis in G1-S state. It also increases expression of N-myc down-regulated gene 1 which can suppress metastasis in cancer. It has been suggested that Iron chelators may decrease leukemic tumor growth in animal models of acute myeloid leukemia (AML). Some other case studies demonstrated the role of Iron chelators in relapse and/or refractory AML. Finally a phase 1 clinical study is undertaken for evaluate the role of Tiapine and cytarabine for adult AML and high-risk myelodysplastic syndrome. So in this study the investigators try to evaluate the role of iron chelating agent (deferasirox) for patients with acute lymphatic leukemia (ALL) and AML patients who cannot be treated with standard chemotherapy regimes .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute leukemia (myeloid or lymphoblastic) who do not receive the standard chemotherapy regimens for treatment; because of the following reasons:

1. age > 65
2. existence of another illness, such as heart failure (EF> 40)

2. Ferritin < 500 μg / l

3. Not existence of other co morbidity

4. GFR > 40

Exclusion Criteria:

1. GFR < 40
2. Control group become iron overloaded (Ferritin > 500 μg /l)
3. Incidence of any severe gastrointestinal symptoms (Mucositis, Enterocolitis, Typhlitis, Nausea, Diarrhea)
4. Not willing to continue treatment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
complete Remission | first month

SECONDARY OUTCOMES:
Partial Remission | up to four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Valiollah Mehrzad, MD, Principal Investigator — Seyyed-alshohada hospital of Isfahan; Shaghayegh Haghjoo Javanmard, MD, PHD, Principal Investigator — Applied Physiology Research Center; Mahnaz Danesh, MD, Principal Investigator — Seyyed-alshohada hospital of Isfahan; Alireza Eishi, Med student, Principal Investigator — Applied Physiology Research Center

REFERENCES:
- [Background] Heath JL, Weiss JM, Lavau CP, Wechsler DS. Iron deprivation in cancer--potential therapeutic implications. Nutrients. 2013 Jul 24;5(8):2836-59. doi: 10.3390/nu5082836. PMID 23887041
- [Background] Paubelle E, Zylbersztejn F, Alkhaeir S, Suarez F, Callens C, Dussiot M, Isnard F, Rubio MT, Damaj G, Gorin NC, Marolleau JP, Monteiro RC, Moura IC, Hermine O. Deferasirox and vitamin D improves overall survival in elderly patients with acute myeloid leukemia after demethylating agents failure. PLoS One. 2013 Jun 20;8(6):e65998. doi: 10.1371/journal.pone.0065998. Print 2013. PMID 23840388
- [Background] Fukushima T, Kawabata H, Nakamura T, Iwao H, Nakajima A, Miki M, Sakai T, Sawaki T, Fujita Y, Tanaka M, Masaki Y, Hirose Y, Umehara H. Iron chelation therapy with deferasirox induced complete remission in a patient with chemotherapy-resistant acute monocytic leukemia. Anticancer Res. 2011 May;31(5):1741-4. PMID 21617233
- See also: Deferasirox Information — http://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafetyInformationforPatientsandProviders/ucm183861.htm